CLINICAL TRIAL: NCT00713167
Title: Randomized, Cross-Over, Double Blind, Placebo-Controlled Study of Grape Seed Extract in Treating Patients With Mild Hyperlipidemia
Brief Title: The Efficacy of Red Grape Seed Extract on Lipid Profile and Oxidized Low-Density Lipoprotein (OX-LDL)
Acronym: GSE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Tabriz University (Other)
Responsible Party: Maryam Keshtkar Jahromi, Shahid Beheshti University (MC)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBMU 87-01-106-5694
Record Dates: First submitted 2008-07-08; First posted 2008-07-11 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Hyperlipidemia
Keywords: Grape Seed Extract; Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grape Seed Extract (Experimental): Enrolled patients who are randomly assigned to receive Grape Seed Extract capsules
  Interventions: Drug: Grape Seed Extract (Vitagrape)
- Placebo (Placebo Comparator): Placebo enrolled patients who are randomly assigned to receive placebo of Grape Seed Extract
  Interventions: Drug: Placebo of Grape Seed Extract

INTERVENTIONS:
Drug: Grape Seed Extract (Vitagrape) — Drug {Each Containing: Grape Seed Extract100 mg +...}
  1 capsule twice daily for 2 months
  Other Names: Vitagrape; Iran Ministry of Health Registration Number: 5/92/43198
  Arms: Grape Seed Extract
Drug: Placebo of Grape Seed Extract — Placebo {Each Containing: Gelatin 17mg + Cellulose Microcrystalline (Avicel) 67 mg + Dicalcium Phosphate 216mg}
  1 capsule twice daily for 2 months
  Arms: Placebo

SUMMARY:
Antioxidants are potent scavengers of free radicals and serve as inhibitors of neoplastic processes. A large number of synthetic and natural antioxidants are known to induce beneficial effects on human health and disease prevention. Cardioprotective ability of grape seed extract polyphenols (GSEP) was studied in animals and humans. It has been suggested that grape seed proanthocyanidins have cardioprotective effects against reperfusion-induced injury of free radicals after ischemia. In another study, it is suggested that proanthocyanidins, the major polyphenols in red wine, might trap reactive oxygen species in aqueous series such as plasma and interstitial fluid of the arterial wall; thereby inhibiting oxidation of low-density lipoprotein (LDL) and showing an antiatherosclerotic activity. The only human model study designed to evaluate the effect of a standardized formulation of a GSEP (leucoselect-phytosome [LP]) on the susceptibility of LDL to oxidation in a group of heavy smokers, revealed that the antioxidant potential of GSEP may be effective in oxidative stress (smoking); however more investigational data are needed before wider use in clinical settings. Based on these observations, the investigators decided to evaluate the effect of GSEP in reducing OX-LDL in patients diagnosed with mild hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Triglyceride > 150 mg/dl
2. Total Cholesterol > 200 mg/dl

Exclusion Criteria:

1. Severe hyperlipidemia (Triglyceride > 300 mg/dl,Total Cholesterol > 250 mg/dl)
2. Usage of antilipid drugs
3. Herbivore Diet
4. Alcoholism
5. Heart failure
6. Known cases of any malignancy
7. BMI > 30 kg/M2
8. Chronic Hepatic Diseases
9. Smoking
10. Chronic Renal Failure

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
OX-LDL | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed

SECONDARY OUTCOMES:
LDL | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed
HDL | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed
Blood Pressure | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed
Triglyceride | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed
Total Cholesterol | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed
Body Mass Index | 8 weeks -{45 days wash out, crossed }- 8 weeks after crossed
LDL/HDL | 8 weeks- {45 days wash out, crossed }- 8 weeks after crossed

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Keshtkar-Jahromi, MD,, Study Director — Shahid Beheshti University (MC); Hassan Argani, MD, Study Chair — Shahid Beheshti University (MC); Abbas Delazar, PhD, Principal Investigator — Tabriz University; Ali Eskandari, MD, Principal Investigator — Shahid Beheshti University (MC); Sharareh Gholamin, MD, Principal Investigator — Shahid Beheshti University (MC); Seyed Mostafa Razavi, MD, Principal Investigator — Shahid Beheshti University (MC)
Locations (2):
- Iran (2):
  - Ghorbanihaghjo, Tabriz, East Azarbayejan
  - Maryam, Tehran, Tehran Province

REFERENCES:
- [Background] Bagchi D, Bagchi M, Stohs SJ, Das DK, Ray SD, Kuszynski CA, Joshi SS, Pruess HG. Free radicals and grape seed proanthocyanidin extract: importance in human health and disease prevention. Toxicology. 2000 Aug 7;148(2-3):187-97. doi: 10.1016/s0300-483x(00)00210-9. PMID 10962138
- [Background] Bagchi D, Sen CK, Ray SD, Das DK, Bagchi M, Preuss HG, Vinson JA. Molecular mechanisms of cardioprotection by a novel grape seed proanthocyanidin extract. Mutat Res. 2003 Feb-Mar;523-524:87-97. doi: 10.1016/s0027-5107(02)00324-x. PMID 12628506
- [Background] Pataki T, Bak I, Kovacs P, Bagchi D, Das DK, Tosaki A. Grape seed proanthocyanidins improved cardiac recovery during reperfusion after ischemia in isolated rat hearts. Am J Clin Nutr. 2002 May;75(5):894-9. doi: 10.1093/ajcn/75.5.894. PMID 11976164
- [Background] Joshi SS, Kuszynski CA, Bagchi D. The cellular and molecular basis of health benefits of grape seed proanthocyanidin extract. Curr Pharm Biotechnol. 2001 Jun;2(2):187-200. doi: 10.2174/1389201013378725. PMID 11480422
- [Background] Bagchi D, Garg A, Krohn RL, Bagchi M, Bagchi DJ, Balmoori J, Stohs SJ. Protective effects of grape seed proanthocyanidins and selected antioxidants against TPA-induced hepatic and brain lipid peroxidation and DNA fragmentation, and peritoneal macrophage activation in mice. Gen Pharmacol. 1998 May;30(5):771-6. doi: 10.1016/s0306-3623(97)00332-7. PMID 9559333
- [Background] Yamakoshi J, Kataoka S, Koga T, Ariga T. Proanthocyanidin-rich extract from grape seeds attenuates the development of aortic atherosclerosis in cholesterol-fed rabbits. Atherosclerosis. 1999 Jan;142(1):139-49. doi: 10.1016/s0021-9150(98)00230-5. PMID 9920515
- [Background] Zhang FL, Gao HQ, Wu JM, Ma YB, You BA, Li BY, Xuan JH. Selective inhibition by grape seed proanthocyanidin extracts of cell adhesion molecule expression induced by advanced glycation end products in endothelial cells. J Cardiovasc Pharmacol. 2006 Aug;48(2):47-53. doi: 10.1097/01.fjc.0000242058.72471.0c. PMID 16954821
- [Background] Vigna GB, Costantini F, Aldini G, Carini M, Catapano A, Schena F, Tangerini A, Zanca R, Bombardelli E, Morazzoni P, Mezzetti A, Fellin R, Maffei Facino R. Effect of a standardized grape seed extract on low-density lipoprotein susceptibility to oxidation in heavy smokers. Metabolism. 2003 Oct;52(10):1250-7. doi: 10.1016/s0026-0495(03)00192-6. PMID 14564675